CLINICAL TRIAL: NCT02871414
Title: REST: Restoring Effective Sleep Tranquility in College Veterans With Service-Related Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Aaron Eakman, Assistant Professor, Colorado State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-5974H
Record Dates: First submitted 2016-08-02; First posted 2016-08-18 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- REST - Early Group (Experimental): Intervention - 7 weeks of sleep skills education provided in group and one-on-one format
  Interventions: Behavioral: REST - Early Group
- REST - Late Group (Experimental): Control - No treatment for 7 weeks, then provided 7 weeks of sleep skills education provided in group and one-on-one format
  Interventions: Behavioral: REST - Late Group

INTERVENTIONS:
Behavioral: REST - Early Group — Intervention - 7 weeks of sleep skills education provided in group and one-on-one format
  Arms: REST - Early Group
Behavioral: REST - Late Group — Control for REST - Early Group, then provided group and one-on-one sleep education and sleep skills intervention
  Arms: REST - Late Group

SUMMARY:
The purpose of the project is to improve the sleep quality and sleep duration of post 9/11 veterans seeking college degrees. Preliminary research findings within CSU's New Start for Student Veterans program indicate veterans with service-related injuries report difficulties with sleep quality and duration. The REST program will recruit 24 college veterans and engage them in a seven-week multi component sleep improvement program using evidence-based educational and behavioral change supports that are considered best practice for improving sleep quality. The investigators' scientific objectives in this application are to establish the efficacy of a group-based sleep education and sleep-skills intervention to improve sleep quality and duration, and to advance understanding of relationships between participants' sleep-related knowledge and behaviors associated with improved sleep quality and duration in veterans with service-related injuries in college. The investigators will initially engage 8 participants to establish treatment fidelity and participant satisfaction of the 7-week group intervention. This will be followed by engaging 16 additional participants in the 7-week group intervention, 8 will be randomly placed as wait-list controls and then receive the intervention. The 7-week group intervention will take place within the CSU Occupational Therapy Department, and all assessments will be completed using a web-based survey.

DETAILED DESCRIPTION:
Design: The investigators will complete a mixed-methods prospective longitudinal study with pre and post intervention testing (component A; N = 8), followed by a mixed-methods wait-listed cross-over controlled trial with pre and post intervention testing (component B; N = 16). Within component A participants will complete pre-intervention assessments, complete 7-weeks of group intervention and weekly monitoring, and complete post-intervention assessments and follow-up assessments 3 months later. Within component B, 8 participants will be randomly assigned to the early intervention group and 8 participants will be assigned to the wait-listed cross-over (or late) intervention group. Participants in the early and late groups will complete pre-intervention assessments at the same time. Participants in the early intervention group will then complete 7-weeks of group intervention and weekly monitoring, and complete post-intervention assessments immediately after the intervention and a follow-up assessment 3 months later. Participants in the late intervention group will complete sleep diary information for 7 randomly-chosen nights, a second pre-intervention assessment approximately 8-weeks following their initial pre-intervention assessment, complete 7-weeks of group intervention and weekly monitoring, and complete post-intervention assessments and follow-up assessments 3 months later. All interventions will occur within the CSU Occupational Therapy Department, all pre and post intervention assessments will be completed using a web-based survey.

Participants: Active recruitment of study participants will occur through email and telephone contacts to veterans engaged in ongoing CSU IRB-approved studies in which they have agreed to being contacted regarding participation in future studies occurring within the Department of Occupational Therapy and the New Start for Student Veterans Program. Participants will receive a gift card of their choice for completing post-intervention assessments, whereas participants assigned to the late group of Component B will receive an additional gift card for completing their second pre-intervention assessment. Participants who complete the 7- week group intervention and first of two post-intervention assessments will also be allowed to keep the Fitbit wearable actigraph they have used within the study.

Data Collection: The investigators will complete a comprehensive evaluation at each assessment period. Data collected will address 2 aims. Aim 1 will assess the fidelity and participant satisfaction of a group-delivered sleep education and sleep skills intervention for veterans with service-related injuries who are in college. The working hypothesis is that a group-delivered sleep education and sleep skills intervention will be safe, demonstrate adequate treatment fidelity, and participant satisfaction. Aim 2 will assess the efficacy of a group-delivered sleep education and sleep skills intervention for veterans with service-related injuries who are in college in terms of key variables of interest. The working hypothesis is that participation in a group-delivered sleep education and sleep skills intervention will result in improvements in participants' sleep quality, sleep duration, and mental health. Further, through the evaluation of program data including participants' attendance, sleep-related knowledge and behaviors, program adherence, and qualitative interview data we seek to understand the key processes and outcomes associated with intervention efficacy. Please see the Outcome Measures section of this protocol registration for name and purpose of outcomes.

Intervention: All post 9/11 veteran participants will complete a 7-week group sleep education and sleep skills intervention within the Department of Occupational Therapy. The investigators will deliver a sleep education and sleep skills group-based intervention based upon established best-practices for improving sleep quality and sleep quantity associated with insomnia, specifically targeted to student veterans with service-related injuries. All components of the intervention will be delivered by registered and licensed occupational therapists practicing within the New Start for Student Veterans Program and the Department of Occupational Therapy, which serves college veterans with service-related injuries at CSU and Front Range Community College. For the duration of the study two local physicians, board certified in Sleep Medicine and Psychiatry respectively will be available for consultation on sleep issues related to veterans. The 7-week group intervention was developed to improve sleep quality and sleep quantity through sleep-related education and behavioral goal setting addressing: sleep monitoring with actigraph and sleep log, sleep education, sleep hygiene and development and maintenance of good sleep habits, stimulus control for sleep preparation, and mindfulness/ yoga for sleep preparation and daily stress reduction. Participants will also meet individually either in person or by telephone on a weekly basis with a registered and licensed occupational therapist, experienced in working with student veterans with service-related injuries, and knowledgeable of the sleep-related education used within the intervention. Individualized meetings will be used to assure: 1) understanding and adherence in the use of sleep monitoring actigraphy and sleep diaries, and 2) establishing and monitoring participants' individualized goals related to sleep skills behaviors. Participants will also have access to an occupational therapist from CSU's Assistive Technology and Resource Center, experienced in working with veterans with service-related injuries, to support the use of Fitbit sleep actigraph and associated mobile sleep applications to ensure understanding of Fitbit use, integration (sync) of Fitbit and mobile application, and establishment of an anonymous web-based profile for monitoring sleep-related data.

Data Analysis: For Aim 1, the investigators will assess the intervention fidelity and participant satisfaction of a group delivered sleep education and sleep skills intervention, the investigators will report proportions of educational content and behavioral goals established, and proportions of participants who rate the interventions as enjoyable (1-4 on Likert scale). Descriptive statistics will be used to examine means and variances of key constructs of interest. Change in key variables over the 7-week intervention will be inspected via individual growth charts. Attendance, attrition, and adverse events will be reported as proportions. The investigators will use focus groups to formally evaluate the program, and to elicit suggestions for program improvement. Importantly, participants will be asked to describe changes that have occurred during the intervention and why they think the sleep education and behavioral sleep goals helped improve sleep quality, sleep quantity or other sleep-related variables, such as mindfulness, physical, mental, and social health domains. Qualitative analytic software (e.g., Atlas TI) will be used to code segments of qualitative data. The investigators will review the text and identify emergent themes and use an iterative consensus building process to generate themes and codes for participants and their spouses/ significant others. For Aim 2 quantitative data will be analyzed in two ways. First, for constructs measured at pre and post intervention only, a repeated-measures ANOVA will be conducted to determine if post-intervention scores differ significantly across the early and delayed conditions. Second, for the sleep variables, which will be collected on a daily basis during the intervention, a time-series approach will be used to examine within person change in these constructs over time. This type of analysis models the effect of an intervention on a meaningful outcome collected regularly over time - with measurements before the implementation of the intervention, during the intervention, and ideally after the intervention. Using time-series models, the effect of an intervention can be estimated after adjusting for serial dependence and any other measured shifts (e.g., day of the week, length of the day, mid-terms/finals, outside temperature), through the specification of linear models that capture increases or decreases in the mean level or slope of the time-series. Specifically, an Auto-regressive Integrated Moving Average (ARIMA) model will be used to examine intervention effects of the program for the identified outcomes.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in university classes
* age 18 or older
* self-report a service-related injury
* present a U.S. Military DD-214 form indicating honorable separation from service
* 10 or higher on the Insomnia Severity Index

Exclusion Criteria:

* Unstable bipolar disorder
* active seizure disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study Sleep Measure | Change from Baseline Medical Outcomes Study Sleep Measure at 7 weeks
  Measuring sleep quality and quantity.
PROMIS Sleep Disturbances Scale (short form) | Change from Baseline PROMIS Sleep Disturbances Scale (short form) at 7 weeks
  Measuring sleep quality and quantity.
Pittsburgh Sleep Quality Index Addendum for PTSD | Change from Baseline Pittsburgh Sleep Quality Index Addendum for PTSD at 7 weeks
  Measuring sleep quality and quantity.
Insomnia Severity Index | Change from Baseline Insomnia Severity Index at 7 weeks
  Measures severity of sleep-onset, sleep maintenance, early morning awakening, satisfaction with current sleep, interference with daily function, noticeability of impairments related to sleep problems, and level of distress caused by sleep problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided